CLINICAL TRIAL: NCT06266715
Title: A Double-blind Randomized Controlled Trial of Adenosine Disodium Triphosphate in Improving Moderate to Severe Depressions
Brief Title: Improvement of Depression With Use of ATP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2024-070
Record Dates: First submitted 2024-01-31; First posted 2024-02-20 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Cap escitalopram 10mg once daily (OD) for four weeks and injection 110ml NS twice daily (BD) for two weeks.
  Interventions: Drug: Placebo Group
- ATP Group (Experimental): Cap escitalopram 10mg OD for four weeks and injection ATP 100mg in 100ml NS BD for two weeks.
  Interventions: Drug: ATP Group

INTERVENTIONS:
Drug: ATP Group — Cap escitalopram 10mg OD for four weeks and injection ATP 100mg in 100ml NS BD for two weeks.
  Arms: ATP Group
Drug: Placebo Group — Cap escitalopram 10mg OD for four weeks and injection110ml NS BD for two weeks.
  Arms: Placebo Group

SUMMARY:
This clinical study is a randomized, double-blind, placebo-controlled trial with an intervention period of 4 weeks. Participants will be patients with moderate to severe depression who meet the inclusion criteria during the screening period. After recruitment written informed consent form will be signed and the baseline evaluation will be done then the treatment period follows. The subjects will be randomly assigned to a control group (escitalopram plus normal saline(NA)) and an ATP group (escitalopram plus adenosine disodium triphosphate(ATP)) in a 1:1 ratio for treatment, with a total number of 120 recruited patients. Assessment will be carried out as an analysis of changes in Hamilton Depression Scale（HAMD-24）, cognitive function test, brain functional network, inflammatory markers, and other indicators in the first, second, and fourth week of intervention which will evaluate the effectiveness of ATP in improving moderate to severe depression preliminarily.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic and statistical manual of mental disorders-5 diagnostic criteria for moderate to severe depression.
* HAMD-24 scores ≥ 20.
* 18-65 female or male.
* Participants who have not used any psychotropic medications within one month prior to study and never had a treatment with escitalopram.
* Individuals without contraindications to selective serotonin reuptake inhibitor.
* Individuals without contraindications to ATP.
* Written informed consent.

Exclusion Criteria:

* Participants with various major mental disorders other than depression (bipolar disorder, any psychotic disorder, Personality Disorders, alcohol use disorder, substance use disorder, and disorders due to medical or organic cause) assessed using Chinese version of the Mini International Neuropsychiatric Interview (MINI).
* Individuals with neurological disorders such as dementia.
* Individuals with a high risk of suicide.
* Pregnant and lactating women.
* Contraindications to MRI.
* Physician evaluation was not suitable for participants in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HAMD-24 | Baseline, two weeks, and four weeks
  Changes in HAMD-24. Score range from 0-76, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Diffusion Tensor Imaging | Baseline, two weeks, and four weeks
  Diffusion Tensor Imaging(DTI) is used to detect changes in fractional anisotropy (FA) maps of brain white matter fiber in major depressive patients.
Diffusion Spectral Imaging | Baseline, two weeks, and four weeks
  Diffusion Spectral Imaging(DSI) is a newly proposed modification of DTI that allows potentially improved visualization of the complex white matter architecture.
Quantitative susceptibility mapping | Baseline, two weeks, and four weeks
  Quantitative susceptibility mapping(QSM) is widely used by the imaging research community in applications to detect iron. Tissue can become magnetized in response to a magnetic field, and the extent of magnetization is known as susceptibility, which arises from unpaired electrons in iron or external sources such as contrast agents. QSM permits visualization of the sizes and shapes of iron sources, delivers precise estimates of iron concentrations (units: parts per billion [ppb] or parts per million [ppm]).
Monetary Incentive Delay Task | Baseline, two weeks, and four weeks
  Participants see cues that they may win or lose money, then wait for a variable anticipatory delay period, and respond to a rapidly presented target with a single button press to try to either win or avoid losing money.
  Task-based functional magnetic resonance imaging (fMRI) will be used to assess neural activity during the Monetary Incentive Delay Task.
Emotional faces processing task | Baseline, two weeks, and four weeks
  Volunteers responded with a button press to each face with different emotions, indicating whether it was male or female.
  Task-based functional magnetic resonance imaging (fMRI) will be used to assess neural activity during the emotional faces processing task.
Resting state functional connectivity | Baseline, two weeks, and four weeks
  Resting-state functional connectivity will be assessed over a 10-minute period, focusing on functional connectivity between the medial prefrontal cortex and Lhb.
Hamilton Anxiety Scale | Baseline, one week, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in Hamilton Anxiety Scale(HAMA-14). Score range from 0-56, higher scores mean a worse outcome.
Clinical Global Impression | Baseline, one week, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in Clinical Global Impression(CGI)
Snaith-Hamilton Pleasure Scale | Baseline, one week, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in Snaith-Hamilton Pleasure Scale(SHAPS). Score range from 14-56, higher scores mean a worse outcome.
Insomnia Severity Index | Baseline, one week, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in Insomnia Severity Index(ISI). Score range from 0-28, higher scores mean a worse outcome.
Columbia-Suicide Severity Rating Scale | Baseline, one week, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in Columbia-Suicide Severity Rating Scale(C-SSRS)
Antidepressants Side Effects | One week, two weeks, four weeks, twelve weeks, twenty-four weeks
  Number of Participants with antidepressants side effects(SERS)
C-reactive protein | Baseline, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in C-reactive protein(CRP)
Tumor Necrosis Factor α | Baseline, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in Tumor Necrosis Factor α(TNF-α)
Interleukin- 6 | Baseline, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in interleukin- 6(IL-6)
N-back task | Baseline, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in reaction time and accuracy
Attention network test | Baseline, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in reaction time and accuracy
Psychomotor vigilance task | Baseline, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in reaction time and accuracy
Hamilton Depression Scale | Baseline, one week, twelve weeks, twenty-four weeks
  Changes in HAMD-24. Score range from 0-76, higher scores mean a worse outcome.
Montgomery and asberg Depression Rating Scale | Baseline, one week, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in Montgomery and asberg (MADRS) Depression Rating Scale. Score range from 0-60, higher scores mean a worse outcome.
Beck Depression Inventory | Baseline, one week, two weeks, four weeks, twelve weeks, twenty-four weeks
  Changes in Beck Depression Inventory(BDI). Score range from 0-63, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xin Q, Wei H, Paudel D, Hu N, Zhao Y, Feng Y, Luo X, Su M, Xue X, Huang H, Lv Z, Tang C, Zhao Y, Tan M, Luo X, Yang Y, Liu Q, Huang M, Cheng Y, Gao T, Zhang B. Intravenous administration of adenosine triphosphate combined with escitalopram in major depressive disorder: protocol for a randomised, double-blind, placebo-controlled trial. BMJ Open. 2025 Aug 28;15(8):e098281. doi: 10.1136/bmjopen-2024-098281. PMID 40876882